CLINICAL TRIAL: NCT00860470
Title: Antenatal Multiple Micronutrient Supplementation to Improve Infant Survival and Health in Bangladesh
Brief Title: Antenatal Micronutrient Supplementation and Infant Survival
Acronym: JiVitA-3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Mahidol University (Other); Johns Hopkins University (Other); Beximco Pharmaceuticals Ltd. (Industry); DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JHU_IRB 570
Record Dates: First submitted 2009-03-11; First posted 2009-03-12 (Estimated); Results first posted 2015-05-27 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Infant Mortality; Preterm Birth; Low Birth Weight; Neonatal Mortality; Perinatal Mortality
Keywords: micronutrients; deficiency; pregnancy; birth outcomes; infant mortality; neonatal mortality; malnutrition; antenatal
MeSH Terms: conditions — Infant Death; Premature Birth; Perinatal Death; Malnutrition | interventions — Iron; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Iron (27 mg) and folic acid (600 ug)
  Interventions: Dietary Supplement: Iron (27 mg) - folic acid (600 ug)
- 2 (Experimental): Multiple micronutrient
  Interventions: Dietary Supplement: Multiple micronutrient

INTERVENTIONS:
Dietary Supplement: Iron (27 mg) - folic acid (600 ug) — Supplement serves as the "Control" (providing the current standard of care during pregnancy). Mothers instructed to take 1 tablet per day, from the 1st trimester through 12 weeks post-partum.
  Other Names: iron-folate
  Arms: 1
Dietary Supplement: Multiple micronutrient — Containing 15 micronutrients all at an RDA including: vitamin A (770 ug retinol equivalents, vitamin D (5 ug), vitamin E (15 mg), folic acid (600 ug), thiamin (1.4 mg), riboflavin (1.4 mg), niacin (18 mg), vitamin B-12 (2.6 mg), vitamin B-6 (1.9 mg), vitamin C (85 mg), iron (27 mg), zinc (12 mg), iodine (220 ug), copper (1000 ug), selenium (60 ug).
  Mothers instructed to take 1 tablet per day, from the 1st trimester through 12 weeks post-partum.
  Other Names: one-a-day multivitamin; antenatal micronutrient
  Arms: 2

SUMMARY:
The purpose of this community-based randomized trial is to examine whether a daily antenatal and postnatal multiple micronutrient supplement given to women will enhance newborn and infant survival and health and other birth outcomes in a rural setting in northwestern Bangladesh.

DETAILED DESCRIPTION:
Maternal deficiency in multiple essential micronutrients is likely to be a major public health problem in low-income countries. Supplementing mothers with certain individual micronutrients has been shown to confer health benefits, although the evidence is not clear for multiple micronutrients. We aim to test, in a cluster-randomized, double-masked, controlled trial whether giving a daily multiple micronutrient supplement (similar in composition to the UNICEF antenatal supplement) will enhance infant survival and birth outcomes such as birth weight and gestational duration in a rural population in Bangladesh. Over the duration of 2-3 years a community-surveillance in the northwestern, rural Districts of Gaibandha and Southern Rangpur, the trial plans to identify and recruit 45,000 pregnant women based on 5-weekly histories of amenorrhea confirmed by urine-testing, and supplement them with either a multiple micronutrient supplement or an iron-folic acid supplement (as the standard of care control for pregnancy) and monitor pregnancy health, birth outcomes and vital status and health of liveborn infants through 6 months of age. In a ~3% sub-sample of mothers, additional measures of nutritional and health status will be evaluated in the 1st and 3rd trimesters of pregnancy, and at 3 months postpartum (with infants), that include anthropometric and body composition (bioelectrical impedance) assessment, collection of biospecimens (eg, phlebotomy and breast milk sampling for micronutrient and other analyte concentration determinations), and other clinical assessments. The trial will generate evidence from which to examine the safety and efficacy of an antenatal through postnatal maternal micronutrient supplement intervention in order to inform and guide antenatal nutrition policies and programs in South Asia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and consents to participate

Exclusion Criteria:

* Not interviewed for consent within 12 consecutive weeks after being ascertained as pregnant by urine testing

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44567 (Actual)
Dates: Start 2008-01; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith P West, Jr., Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Parul Christian, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States
- JiVitA Project Office, Rangpur City, Gaibandha District, Bangladesh

REFERENCES:
- [Background] Christian P, Khatry SK, Katz J, Pradhan EK, LeClerq SC, Shrestha SR, Adhikari RK, Sommer A, West KP Jr. Effects of alternative maternal micronutrient supplements on low birth weight in rural Nepal: double blind randomised community trial. BMJ. 2003 Mar 15;326(7389):571. doi: 10.1136/bmj.326.7389.571. PMID 12637400
- [Background] Christian P. Micronutrients and reproductive health issues: an international perspective. J Nutr. 2003 Jun;133(6):1969S-1973S. doi: 10.1093/jn/133.6.1969S. PMID 12771347
- [Background] Christian P, Shrestha J, LeClerq SC, Khatry SK, Jiang T, Wagner T, Katz J, West KP Jr. Supplementation with micronutrients in addition to iron and folic acid does not further improve the hematologic status of pregnant women in rural Nepal. J Nutr. 2003 Nov;133(11):3492-8. doi: 10.1093/jn/133.11.3492. PMID 14608063
- [Background] Christian P, West KP, Khatry SK, Leclerq SC, Pradhan EK, Katz J, Shrestha SR, Sommer A. Effects of maternal micronutrient supplementation on fetal loss and infant mortality: a cluster-randomized trial in Nepal. Am J Clin Nutr. 2003 Dec;78(6):1194-202. doi: 10.1093/ajcn/78.6.1194. PMID 14668283
- [Background] Katz J, West KP Jr, Khatry SK, Christian P, LeClerq SC, Pradhan EK, Shrestha SR. Risk factors for early infant mortality in Sarlahi district, Nepal. Bull World Health Organ. 2003;81(10):717-25. Epub 2003 Nov 25. PMID 14758431
- [Background] Jiang T, Christian P, Khatry SK, Wu L, West KP Jr. Micronutrient deficiencies in early pregnancy are common, concurrent, and vary by season among rural Nepali pregnant women. J Nutr. 2005 May;135(5):1106-12. doi: 10.1093/jn/135.5.1106. PMID 15867289
- [Background] Christian P, Osrin D, Manandhar DS, Khatry SK, de L Costello AM, West KP Jr. Antenatal micronutrient supplements in Nepal. Lancet. 2005 Aug 27-Sep 2;366(9487):711-2. doi: 10.1016/S0140-6736(05)67166-8. No abstract available. PMID 16125578
- [Background] Christian P, Jiang T, Khatry SK, LeClerq SC, Shrestha SR, West KP Jr. Antenatal supplementation with micronutrients and biochemical indicators of status and subclinical infection in rural Nepal. Am J Clin Nutr. 2006 Apr;83(4):788-94. doi: 10.1093/ajcn/83.4.788. PMID 16600929
- [Background] Katz J, Christian P, Dominici F, Zeger SL. Treatment effects of maternal micronutrient supplementation vary by percentiles of the birth weight distribution in rural Nepal. J Nutr. 2006 May;136(5):1389-94. doi: 10.1093/jn/136.5.1389. PMID 16614435
- [Background] West KP Jr, Christian P. Antenatal micronutrients in undernourished people. Lancet. 2008 Feb 9;371(9611):452-4. doi: 10.1016/S0140-6736(08)60214-7. No abstract available. PMID 18262025
- [Background] Christian P, Darmstadt GL, Wu L, Khatry SK, Leclerq SC, Katz J, West KP Jr, Adhikari RK. The effect of maternal micronutrient supplementation on early neonatal morbidity in rural Nepal: a randomised, controlled, community trial. Arch Dis Child. 2008 Aug;93(8):660-4. doi: 10.1136/adc.2006.114009. PMID 18644934
- [Background] Shankar AH, Genton B, Baisor M, Paino J, Tamja S, Adiguma T, Wu L, Rare L, Bannon D, Tielsch JM, West KP Jr, Alpers MP. The influence of zinc supplementation on morbidity due to Plasmodium falciparum: a randomized trial in preschool children in Papua New Guinea. Am J Trop Med Hyg. 2000 Jun;62(6):663-9. doi: 10.4269/ajtmh.2000.62.663. PMID 11304051
- [Derived] de Boer M, Thorne-Lyman AL, Shamim AA, Wu LS, Shaikh S, Ali H, West KP, Christian P. Dietary diversity as a modifier of the effect of supplementation with multiple micronutrients during pregnancy on low birth weight in a randomized controlled trial in Bangladesh. Am J Clin Nutr. 2025 Sep;122(3):762-769. doi: 10.1016/j.ajcnut.2025.07.007. Epub 2025 Jul 12. PMID 40653272
- [Derived] Finkelstein JL, Cuthbert A, Weeks J, Venkatramanan S, Larvie DY, De-Regil LM, Garcia-Casal MN. Daily oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2024 Aug 15;8(8):CD004736. doi: 10.1002/14651858.CD004736.pub6. PMID 39145520
- [Derived] Smith JW, Matchado AJ, Wu LS, Arnold CD, Burke SM, Maleta KM, Ashorn P, Stewart CP, Shaikh S, Ali H, Labrique AB, West KP Jr, Christian P, Dewey KG, Groopman JD, Schulze KJ. Longitudinal Assessment of Prenatal, Perinatal, and Early-Life Aflatoxin B1 Exposure in 828 Mother-Child Dyads from Bangladesh and Malawi. Curr Dev Nutr. 2022 Jan 7;6(2):nzab153. doi: 10.1093/cdn/nzab153. eCollection 2022 Feb. PMID 35155983
- [Derived] Schulze KJ, Gernand AD, Khan AZ, Wu LS, Mehra S, Shaikh S, Ali H, Shamim AA, Sungpuag P, Udomkesmalee E, Labrique AB, West KP, Christian P. Newborn micronutrient status biomarkers in a cluster-randomized trial of antenatal multiple micronutrient compared with iron folic acid supplementation in rural Bangladesh. Am J Clin Nutr. 2020 Nov 11;112(5):1328-1337. doi: 10.1093/ajcn/nqaa223. PMID 32844185
- [Derived] Schulze KJ, Mehra S, Shaikh S, Ali H, Shamim AA, Wu LS, Mitra M, Arguello MA, Kmush B, Sungpuag P, Udomkesmelee E, Merrill R, Klemm RDW, Ullah B, Labrique AB, West KP, Christian P. Antenatal Multiple Micronutrient Supplementation Compared to Iron-Folic Acid Affects Micronutrient Status but Does Not Eliminate Deficiencies in a Randomized Controlled Trial Among Pregnant Women of Rural Bangladesh. J Nutr. 2019 Jul 1;149(7):1260-1270. doi: 10.1093/jn/nxz046. PMID 31006806
- [Derived] Gernand AD, Paul RR, Ullah B, Taher MA, Witter FR, Wu L, Labrique AB, West KP Jr, Christian P. A home calendar and recall method of last menstrual period for estimating gestational age in rural Bangladesh: a validation study. J Health Popul Nutr. 2016 Oct 21;35(1):34. doi: 10.1186/s41043-016-0072-y. PMID 27769295
- [Derived] Christian P, Kim J, Mehra S, Shaikh S, Ali H, Shamim AA, Wu L, Klemm R, Labrique AB, West KP Jr. Effects of prenatal multiple micronutrient supplementation on growth and cognition through 2 y of age in rural Bangladesh: the JiVitA-3 Trial. Am J Clin Nutr. 2016 Oct;104(4):1175-1182. doi: 10.3945/ajcn.116.135178. Epub 2016 Sep 7. PMID 27604769
- [Derived] Gernand AD, Schulze KJ, Nanayakkara-Bind A, Arguello M, Shamim AA, Ali H, Wu L, West KP Jr, Christian P. Effects of Prenatal Multiple Micronutrient Supplementation on Fetal Growth Factors: A Cluster-Randomized, Controlled Trial in Rural Bangladesh. PLoS One. 2015 Oct 2;10(10):e0137269. doi: 10.1371/journal.pone.0137269. eCollection 2015. PMID 26431336
- [Derived] Heaney CD, Kmush B, Navas-Acien A, Francesconi K, Gossler W, Schulze K, Fairweather D, Mehra S, Nelson KE, Klein SL, Li W, Ali H, Shaikh S, Merrill RD, Wu L, West KP Jr, Christian P, Labrique AB. Arsenic exposure and hepatitis E virus infection during pregnancy. Environ Res. 2015 Oct;142:273-80. doi: 10.1016/j.envres.2015.07.004. Epub 2015 Jul 15. PMID 26186135
- [Derived] Sikder SS, Labrique AB, Craig IM, Wakil MA, Shamim AA, Ali H, Mehra S, Wu L, Shaikh S, West KP Jr, Christian P. Patterns and determinants of care seeking for obstetric complications in rural northwest Bangladesh: analysis from a prospective cohort study. BMC Health Serv Res. 2015 Apr 18;15:166. doi: 10.1186/s12913-015-0832-1. PMID 25985774
- [Derived] West KP Jr, Shamim AA, Mehra S, Labrique AB, Ali H, Shaikh S, Klemm RD, Wu LS, Mitra M, Haque R, Hanif AA, Massie AB, Merrill RD, Schulze KJ, Christian P. Effect of maternal multiple micronutrient vs iron-folic acid supplementation on infant mortality and adverse birth outcomes in rural Bangladesh: the JiVitA-3 randomized trial. JAMA. 2014 Dec 24-31;312(24):2649-58. doi: 10.1001/jama.2014.16819. PMID 25536256

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enumeration of women began in December 2007, and active recruitment of pregnant women into the trail began in January 2008. Women were enrolled into the trial by community workers from the projects who visited them at home.
Groups:
- Iron and Folate: Iron (27 mg) and folic acid (600 ug)
  Iron (27 mg) - folic acid (600 ug): Supplement serves as the "Control" (providing the current standard of care during pregnancy). Mothers instructed to take 1 tablet per day, from the 1st trimester through 12 weeks post-partum.
Period: Overall Study
Arm/Group | Iron and Folate | Multiple Micronutrient
Started | 22162 | 22405
Completed | 22114 | 22346
Not Completed | 48 | 59
Not completed — Death | 6 | 10
Not completed — Moved away | 8 | 10
Not completed — Lost to Follow-up | 34 | 39

BASELINE CHARACTERISTICS:
Groups:
- Multiple Micronutrient: Multiple micronutrient
  Multiple micronutrient: Containing 15 micronutrients all at an RDA including: vitamin A (770 ug retinol equivalents, vitamin D (5 ug), vitamin E (15 mg), folic acid (600 ug), thiamin (1.4 mg), riboflavin (1.4 mg), niacin (18 mg), vitamin B-12 (2.6 mg), vitamin B-6 (1.9 mg), vitamin C (85 mg), iron (27 mg), zinc (12 mg), iodine (220 ug), copper (1000 ug), selenium (60 ug).
  Mothers instructed to take 1 tablet per day, from the 1st trimester through 12 weeks post-partum.
- Total: Total of all reporting groups
Arm/Group | Iron and Folate | Multiple Micronutrient | Total
Number analyzed (Participants) | 22,162 | 22,405 | 44567
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (6.43) | 24.4 (6.44) | 24.3 (6.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22,162 | 22,405 | 44567
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian, Bangladeshi | 22,162 | 22,405 | 44567
Region of Enrollment [Number; unit: participants]
  Bangladesh | 22,162 | 22,405 | 44567
Gestational Age in weeks [Mean (Standard Deviation); unit: weeks] | 10.34 (4.7) | 10.28 (4.7) | 10.30 (4.7)
Literacy [Number; unit: participants]
  Literate | 12,816 | 12,985 | 25801
  Illiterate | 9,346 | 9,420 | 18766
Parity [Number; unit: participants with reported data] — Reported for participants for whom baseline data for parity was available
  participants with reported data
    0 | 6,671 | 6,647 | 13318
    1-3 | 13,255 | 13,520 | 26775
    >=4 | 2,186 | 2,194 | 4380
Previous Pregnancy Loss [Number; unit: participants] | 4,974 | 5,106 | 10080

OUTCOME MEASURES:

1. Primary Outcome: Infant Mortality Through 6 mo of Age
Description: Infant Mortality to Age 6 months (180 days from birth)
Time Frame: 6-months post-birth
Population: Not all women recruited into the trial had pregnancies yielding live births. This represents all live births by arm.
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 14142 | 14374
participants | 764 | 741
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p = 0.36, Regression, Logistic; Bonferroni-adjusted alpha=0.01 (for 5 comparisons); Risk Ratio (RR) = 0.95, 95% CI 2-sided [0.86 to 1.06] — GEE with log link function and exchangeable correlation was used to adjust confidence intervals for cluster randomised design; the iron-folic acid supplemented group was the referent

2. Secondary Outcome: Neonatal Mortality
Description: Neonatal Mortality (28 days of life)
Time Frame: 1 month post-birth
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 14142 | 14374
participants | 625 | 626
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p = 0.78, Regression, Logistic; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.88 to 1.20] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Post-neonatal Mortality
Description: Risk of Post-neonatal Mortality (29th -180th day of life)
Time Frame: 1-6 months post-birth
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 13517 | 13748
participants | 139 | 115
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p = 0.11, Regression, Logistic; Risk Ratio (RR) = 0.81, 95% CI 2-sided [0.63 to 1.04] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Still Birth Rates
Description: Stillbirth (born >=24 weeks without breathing, crying, or moving limbs).
Time Frame: 24 weeks gestation to delivery
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 14858 | 15022
participants | 716 | 648
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p = 0.02, Regression, Logistic; Bonferroni-adjusted alpha=0.01 (for 5 comparisons); Risk Ratio (RR) = 0.89, 95% CI 2-sided [0.81 to 0.99] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Preterm Birth
Description: Being born before 37 weeks of gestation
Time Frame: Up to 37 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 13333 | 13475
participants | 2912 | 2510
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Bonferroni-adjusted alpha=0.01 (for 5 comparisons); Risk Ratio (RR) = 0.85, 95% CI 2-sided [0.80 to 0.91] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Extremely Pre-term
Description: Birth before 28 weeks gestation
Time Frame: Up to 28 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 13333 | 13475
participants | 136 | 106
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p = 0.03, Regression, Logistic; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.57 to 0.97] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Very Pre-term
Description: Birth between 28 and 32 weeks of gestation
Time Frame: Between 27 and 33 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 13333 | 13475
participants | 385 | 291
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.62 to 0.86] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Moderate to Late Preterm
Description: Birth between 32 and 37 weeks gestation
Time Frame: Between 31 and 38 weeks of gestation
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 13333 | 13475
participants | 2391 | 2113
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p = 0.87, Regression, Logistic; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.81 to 0.93] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Low Birth Weight
Description: Birth weight below 2500g
Time Frame: Measured at delivery/birth
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 10530 | 10642
participants | 4809 | 4275
Statistical Analysis 1: Comparison: Iron and Folate vs Multiple Micronutrient; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Bonferroni-adjusted alpha=0.01 (for 5 comparisons); Risk Ratio (RR) = 0.88, 95% CI 2-sided [0.85 to 0.91] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Small for Gestation Age
Description: Small for Gestational Age defined as birth weight <10th percentile of a standard reference (Alexander GR, Himes JH, Kaufman RB, et al. Obstet Gynecol. 1996;87(2):163-68).
Time Frame: At delivery/birth
Measure: Number; unit: participants
Arm/Group | Iron and Folate | Multiple Micronutrient
Number analyzed (Participants) | 10099 | 10161
participants | 6479 | 6405
Statistical Analysis 1: Comparison: Iron and Folate; Test type: Superiority or Other; p = 0.13, Regression, Logistic; Bonferroni-adjusted alpha=0.01 (for 5 comparisons); Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.96 to 1.01] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Groups:
- Iron (27 mg) and Folic Acid (600 ug): Iron (27 mg) and folic acid (600 ug)
  Iron (27 mg) - folic acid (600 ug): Supplement serves as the "Control" (providing the current standard of care during pregnancy). Mothers instructed to take 1 tablet per day, from the 1st trimester through 12 weeks post-partum.
Arm/Group | Iron (27 mg) and Folic Acid (600 ug) | Multiple Micronutrient
Serious Adverse Events (participants affected / at risk) | 0/22114 | 0/22346
Other Adverse Events (participants affected / at risk) | 0/22114 | 0/22346

LIMITATIONS AND CAVEATS:
The study was run in an area where iron deficiency rates were low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No